CLINICAL TRIAL: NCT07111143
Title: Empowering Asthmatic Seniors: Nursing Interventions to Mitigate Climate Change-related Effects on Symptom Severity and Physical Capacity
Brief Title: Nursing Interventions to Mitigate Climate Change-related Effects on Symptom Severity and Physical Capacity
Acronym: climate effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norther Private Collage of Nursing (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Amal, Associate professor, researcher, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: senior asthma
Record Dates: First submitted 2025-07-18; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Asthma Exacerbations
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: the study divided into study and control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo, bronchodilator, cortisone if necessary (Sham Comparator): Active comparator: asthmatic medication only
  Interventions: Other: nursing intervention
- education group (Experimental): The intervention group received a nursing intervention, which included three educational sessions classified into one session for the theoretical part through using face to face lecture, discussion, and two sessions for the practical part by utilizing PowerPoint, discussion, demonstration and re-demonstration. The researchers divided the participants into small groups each group consisted 3-4 cases, and three educational sessions provided for each group after data collection.
  Interventions: Other: nursing intervention

INTERVENTIONS:
Other: nursing intervention — medication only

SUMMARY:
Randomize controlled, parallel, double-blind, with two arms, which purpose is verify the nursing educational intervention effects to reduce asthma severity symptoms in older adults.

DETAILED DESCRIPTION:
Climate change is a global concern with far, impacting numerous aspects of human health and well-being especially asthmatic older adults. So that the aim of this study was to evaluate the risk of dry eyes and effectiveness of nursing interventions for reducing climate changes effects on symptoms severity and physical capacity among asthmatic older adults through education to reduce climate effects compared to control group who receive asthma drugs only. This study is a randomize control trail to determine the best care for reducing the severity of symptoms and improve physical capacity from the period from 1/11/ 2024 until 30/4/ 2025. The expected result is decreasing severity of asthma and improve physical capacity.

ELIGIBILITY:
Inclusion Criteria:

* Typically involve confirmation of an asthma diagnosis by a physician
* Age range (often 60 and above ).
* Must be able to provide informed consent and communicate.

Exclusion Criteria:

* Severe comorbidities, recent asthma exacerbations requiring oral corticosteroids
* Inability to communicate effectively or perform necessary lung function tests.
* Cognitive impairments

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
asthma severity | thee month
  Education intervention for asthma prevention. self-management practices and adaptation behaviors: rinsing the nose with salty water, inhalation of steam, proper technique of using inhalers, breathing and Aerobic exercises. Lara Asthma Symptom Scale was used total score between 8 and 40, where higher scores indicate more severe asthma symptoms.

SECONDARY OUTCOMES:
physical activity level among participants | three month
  Education intervention to improv physical capacity. self-management practices and adaptation behaviors: rinsing the nose with salty water, inhalation of steam, proper technique of using inhalers, breathing and Aerobic exercises. International Physical Activity Questionnaire - Short Form adopted is a self-reported tool, in which physical activity grades over the previous seven days were explored and conveyed in metabolic equivalents. The scores for diverse activities were then collected to develop the overall MET-min/week. The physical activity (PA) level was divided into three categories: low (less than 600 MET/min/week), moderate (more than 600 MET/min/week), and high (more than 3000 MET/min/week).

CONTACTS AND LOCATIONS:
Locations (1):
- Norther Private Colleague of Nursing, Arar, Norther Border, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The impact of climate change on the environment, biosphere, and biodiversity has become more evident in the recent years. Human activities have increased atmospheric concentrations of carbon dioxide (CO2 ) and other greenhouse gases. Change in climate an — https://pubmed.ncbi.nlm.nih.gov/32589303/
- Available data/document: Health-Damaging Climate Events Highlight the Need for Interdisciplinary, Engaged Research — https://pubmed.ncbi.nlm.nih.gov/38371354/